CLINICAL TRIAL: NCT05683600
Title: A Multicentre, Randomized, Double-blinded, Placebo-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 as Booster Vaccination in Adults 18 Years of Age or Older
Brief Title: Efficacy and Safety of COVID-19 Vaccine as Booster Vaccination in Adults 18 Years of Age or Older
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: According to the development of the novel coronavirus epidemic situation and the company's R&D decision
Sponsor: Guangzhou Patronus Biotech Co., Ltd. (Industry)
Collaborators: Yantai Patronus Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LYB001/CT-CHN-302
Record Dates: First submitted 2022-12-25; First posted 2023-01-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LYB001 Booster Group (Experimental): Subjects 18 years of age or older who has completed two or three-dose inactivated COVID-19 will receive 30μg LYB001 at day 0 as a booster vaccination.
  Interventions: Biological: Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001
- Placebo Booster Group (Active Comparator): Subjects 18 years of age or older who has completed two or three-dose inactivated COVID-19 will receive placebo at day 0 as a booster vaccination
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 — Intramuscular injection of Recombinant SARS-CoV-2 Vaccine (CHO Cell) LYB001 in the deltoid muscle of the upper arm at day 0. The inoculation dose is 0.5 mL.
  Arms: LYB001 Booster Group
Biological: Placebo — Intramuscular injection of placebo in the deltoid muscle of the upper arm at day 0. The inoculation dose is 0.5 mL.
  Arms: Placebo Booster Group

SUMMARY:
This is an international multicenter clinical trial, which is planned to be conducted in several research centers in China and Pakistan. A randomized, double-blind, placebo-controlled design will be conducted to evaluate the efficacy, safety of LYB001 against COVID-19 as a booster dose in China.

DETAILED DESCRIPTION:
3000 subjects aged 18 years and older who have completed two or three doses of SARS-CoV-2 inactivated vaccine 6-18 months will be enrolled in China. Participants are randomly assigned to LYB001 or placebo group at a ratio of 1:1 and receive one dose at day 0.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18 years and older, including both males and females;
* Subjects who agree to participate in this clinical trial voluntarily and sign the informed consent form, are capable of providing valid identification, understanding and complying with the requirements of the clinical protocol.
* Subjects who have been vaccinated with two-dose or three-dose inactivated COVID-19 vaccine for 6-18 months (including boundary values).
* For female participants of childbearing potential, effective contraception measures should be used within 2 weeks prior to participation in this study and the results of pregnancy test is required to be negative. Participants should voluntarily agree to use effective contraceptive measures from the time of signing the informed consent form to the end of the study (effective contraceptive measures including oral contraceptives (excluding emergency contraceptives), injectable or implantable contraceptives, sustained-release topical contraceptives, hormonal patches, intrauterine device, sterilization, abstinence, condoms (for males), diaphragms, cervical caps, etc.).

Exclusion Criteria:

* Receipt of any COVID-19 vaccines other than inactivated COVID-19 vaccine;
* Systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg (for subjects with poorly controlled blood pressure);
* Axillary body temperature ≥ 37.3°C prior to enrolment;
* Known allergy, or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients;
* History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (MERS);
* History of COVID-19, or positive results for SARS-CoV-2 nucleic acid or antigen tests at screening;
* Receipt of any live attenuated vaccine within 28 days prior to vaccination, and other vaccines such as subunit and inactivated vaccine within 14 days prior to vaccination;
* Receipt of blood or blood-related products, including immunoglobulins, monoclonal antibodies, within 3 months prior to vaccination; or any planned use during the study period.
* Subjects with the following diseases:

  1. Any acute diseases or acute attacks of chronic diseases within 7 days prior to enrolment；
  2. Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.；
  3. Congenital or acquired immunodeficiency or autoimmune disease, or long-term receipt (>14 consecutive days) of glucocorticoid (reference value for dose: ≥20 mg/day prednisone or equivalent) or other immunosuppressive agents within the past 6 months, with exception of inhaled or topical steroids, or short-term use (≤14 consecutive days) of oral corticosteroids；
  4. Currently suffering from or diagnosed with infectious diseases, such as hepatitis B, hepatitis C, syphilis, AIDS etc.；
  5. History or family history of neurological disorders (convulsions, epilepsy, encephalopathy, etc.) or psychiatric disorders；
  6. Asplenia, or functional asplenia；
  7. Presence of severe, uncontrollable or hospitalized cardiovascular diseases, endocrine diseases, blood and lymphatic diseases, immune diseases, liver and kidney diseases, respiratory diseases, metabolic and skeletal diseases, or malignant tumors;
  8. Contraindications to IM injections and blood draws, such as coagulation disorders, thrombotic or bleeding disorders, or conditions that needs continuous anticoagulant usage.
* Drug or alcohol abuse (alcohol intake ≥ 14 units per week) which in the investigator's opinion would compromise the participant's safety or compliance with the study procedures;
* Pregnant or lactating females;
* Having participated or participating in COVID-19 related clinical trials, and those participating or planning to participate in other clinical trials during the study period;
* Presence of any underlying disease or condition which, in the opinion of the investigator, may place the subject at unacceptable risk, is unable to meet the requirements of the protocol, or interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
First occurrence of confirmed symptomatic COVID-19 incidence rate per person-years of follow-up | From 14 days after the booster dose
  First occurrence of confirmed symptomatic COVID-19 incidence rate from 14 days after the booster dose per person-years of follow-up;

SECONDARY OUTCOMES:
The occurrence of adverse events | The occurrence of adverse events within 30 mins,7 days and 28 days after each vaccination
  The occurrence of adverse events within 30 mins,7 days and 28 days after each vaccination
The occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs) | Day 0 to 12 months after vaccination
  The occurrence of serious adverse events (SAEs) and adverse events of special interest (AESIs) within 12 months after vaccination
First occurrence of confirmed severe, critical, and fatal COVID-19 incidence per person-years of follow-up | From 14 days after the booster
  First occurrence of confirmed severe, critical, and fatal COVID-19 incidence from 14 days after the booster dose per person-years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Chengyong Tang, Principal Investigator — Chongqing Bishan District People's Hospital; Li Zhang, Principal Investigator — Shandong Provincial Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Bishan District People's Hospital,Chongqing, Chongqing, Chongqing Municipality
  - Shandong Provincial Center for Disease Control and Prevention, Jinan, Shandong